CLINICAL TRIAL: NCT05770180
Title: A Single-center, Randomized, Double-blind, Controlled Clinical Trial to Evaluate the Safety and Immunogenicity of Booster Vaccination of Recombinant COVID-19 Variant Vaccine (Sf9 Cell) in Healthy People Aged 18 Years and Older
Brief Title: Phase II Clinical Trial of Recombinant COVID-19 Variant Vaccine (Sf9 Cell)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: WestVac Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WSKCT002
Record Dates: First submitted 2023-03-10; First posted 2023-03-15 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low dose test group (Experimental): one dose, Day 0
  Interventions: Biological: Recombinant COVID-19 variant vaccine (Sf9 cell)
- high dose test group (Experimental): one dose, Day 0
  Interventions: Biological: Recombinant COVID-19 variant vaccine (Sf9 cell)
- control group 1 (Active Comparator): one dose, Day 0
  Interventions: Biological: Recombinant COVID-19 vaccine (CHO cell)
- control group 2 (Active Comparator): one dose, Day 0
  Interventions: Biological: Recombinant COVID-19 vaccine (Sf9 cell)

INTERVENTIONS:
Biological: Recombinant COVID-19 variant vaccine (Sf9 cell) — WSK-V102
  Arms: high dose test group; low dose test group
Biological: Recombinant COVID-19 vaccine (CHO cell) — control 1
  Arms: control group 1
Biological: Recombinant COVID-19 vaccine (Sf9 cell) — control 2
  Arms: control group 2

SUMMARY:
A single-center, randomized, double-blind, controlled clinical trial to evaluate the safety and immunogenicity of booster vaccination of Recombinant COVID-19 variant vaccine (Sf9 cell) in healthy people aged 18 years and older after completing 2 or 3 doses of novel coronavirus inactivated vaccine (Vero cells)

DETAILED DESCRIPTION:
two dose level of Recombinant COVID-19 variant vaccine (Sf9 cell) compete with Recombinant COVID-19 vaccine (CHO cell) and Recombinant COVID-19 vaccine (Sf9 cell) .

ELIGIBILITY:
Inclusion Criteria:

1. At the age of 18 or above, consent to participate in the study by voluntarily signing an ICF approved by the Ethics Committee prior to the commencement of any study procedure;
2. Subjects qualified for immunization with this product after medical history, physical examination and clinical judgment of health;
3. Completion of 2 /3 doses of inactivated novel coronavirus vaccine ≥3 months;
4. The subject is able and willing to comply with the requirements of the clinical trial protocol and can complete the study follow-up for approximately 12 months;
5. Armpit body temperature < 37.3℃;
6. Female non-pregnancy period (pregnancy test results are negative), non-lactation period;
7. Fertile women (WOCBP) subjects had taken effective contraceptive measures 1 month before enrollment;
8. WOCBP subjects and male subjects have no pregnancy plans from the screening period to 6 months after the last dose of immunization, and agree to take effective contraceptive measures from the screening visit to 6 months after the last dose of immunization;
9. WOCBP subjects and male subjects agree not to donate eggs (oocytes, oocytes) for assisted reproduction (WOCBP subjects) or to refrain from sperm donation (male subjects) for a period of 6 months from screening visit to the last dose of immunization.

Exclusion Criteria:

1. Positive results of SARS-CoV-2 RT-PCR within 24 hours;
2. The subject has a history of SARS-CoV-2 infection within 3 months;
3. The anti-SARS-CoV-2 IgM antibody was positive during the screening period.
4. History of human coronavirus infection or disease with severe acute respiratory syndrome (SARS), Middle East Respiratory Syndrome (MERS), etc.;
5. Previous history of convulsion, epilepsy, encephalopathy or psychosis or family history;
6. Needle fainter;
7. Those who plan to become pregnant or donate sperm or eggs during the trial period (within 6 months after exemption);
8. Previous history of allergic reaction or allergic reaction to any vaccine and its excipients, such as allergy, urticaria, severe eczema, dyspnea, laryngeal edema, angioneurotic edema, etc.;
9. Received subunit or inactivated vaccine within 14 days or live attenuated vaccine within 1 month prior to receiving the experimental vaccine;
10. Participating in any other interventional test device or drug study within 30 days prior to screening, or currently using another investigational drug or within 5 half-life after the last administration of the study drug;
11. A genetic tendency to hemorrhage or coagulation abnormalities (such as cytokine defects, coagulation disorders or platelet disorders), or a history of severe bleeding, or a history of excessive bleeding or ecchymosis following intramuscular injection or venipuncture;
12. Confirmation of diseases affecting the functioning of the immune system, including cancer, congenital or acquired immunodeficiency (e.g., human immunodeficiency virus (HIV) infection), uncontrolled autoimmune diseases, based on known medical history or diagnosis;
13. There are serious or uncontrollable respiratory diseases, cardiovascular diseases, nervous system diseases, blood and lymphatic system diseases, liver and kidney diseases, metabolic and skeletal system diseases that affect the evaluation of the results of this study as determined by the researchers;
14. Anplenia or functional anplenia;
15. Long-term use (continuous use ≥14 days) of immunosuppressants or other immunomodulatory drugs (such as corticosteroids: prednisone or similar drugs) within the 6 months prior to the study vaccine, but topical use (such as ointment, eye drops, inhalants or nasal spray) is permitted, and the topical use shall not exceed the dosage recommended in the instructions or any systemic signs of exposure;
16. Received immunoglobulin and/or blood products in the three months prior to receiving the study vaccine;
17. Patients undergoing anti-tuberculosis treatment;
18. Medical, psychological, social or other conditions that, in the investigator's judgment, are inconsistent with the protocol or affect the subject's signing of informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
solicited adverse events (AE) | within 14 days after vaccination
  Incidence of solicited adverse events (AE) within 14 days after vaccination
Primary Immunogenic indicator | 14 days after vaccination
  Geometric Mean Titer (GMT) of neutralizing Antibodies against SARS-CoV-2 Prototype and Omicron Variant 14 days after vaccination

SECONDARY OUTCOMES:
unsolicited adverse events | 0-30 days after vaccination
  Incidence of unsolicited adverse events (AE) 0-30 days after vaccination
SAE | within 12 months after vaccination
  Incidence of serious adverse events (SAE), adverse events of Special Concern (AESI), and adverse events requiring medical attention (MAAE) within 12 months after vaccination
GMT | 30 days, 3 months and 6 months after vaccination
  Geometric mean Titer (GMT) of neutralizing Antibodies against SARS-CoV-2 prototype Strain and Omicron Variant Strain
GMI | 14, day 30, 3 and 6 months after vaccination
  Geometric mean growth multiple (GMI) of neutralizing antibody against SARS-CoV-2 prototype strain
binding antibodies | 14, day 30, 3 and 6 months after vaccination
  Geometric Mean Titer (GMT) and Geometric mean Titer Increase Factor (GMI) of IgG Antibody against SARS-CoV-2 S-RBD protein

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial Center for Disease Prevention and Control, Nanjing, China

IPD SHARING:
Plan to Share IPD: No